CLINICAL TRIAL: NCT01556425
Title: The Separate and Combined Effects of Vivitrol and Opiate Abstinence Reinforcement in the Treatment of Opioid Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00052254; 2R01DA019497-06 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-16 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Opioid Dependence
Keywords: opioid use disorder; treatment; heroin; extended-release naltrexone; incentives; cotningency management; employment-based reinforcement; therapeutic workplace
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vivitrol Only (Experimental): The VIVITROL group will be offered one injection of VIVITROL every 4 weeks. Participants in the VIVITROL group will be required to take their scheduled injections to work and earn wages. If a participant misses a scheduled VIVITROL injection (more than 3 days from the scheduled date of administration), the participant will not be allowed to work until the injection is accepted. Additionally, missing a scheduled injection will result in a base pay reset from $8 per hour to $1 per hour. After the reset, the participant's base pay will increase by $1/hour to the maximum of $8/hour for every day that the participant works at least 5 minutes.
  Interventions: Drug: Vivitrol
- VIVITROL&Opiate Abstinence Reinforcement (Experimental): This group will be offered VIVITROL and will be required to take it to attend the workplace and to maintain maximum pay. This group will also receive employment-based opiate abstinence reinforcement. This contingency will require participants to provide opiate-negative urine samples on M,W, and F to maintain their maximum pay. If a participant in this group provides an opiate-positive urine sample, or fails to provide a scheduled sample, their base pay will be reset from $8 per hour to $1 per hour. On each day after the reset that the participant provides a urine sample that meets the opiate abstinence criteria and attends the workplace for at least 5 minutes, their base pay will increase by $1 per hour until it reaches the maximum of $8 per hour.
  Interventions: Drug: Vivitrol; Behavioral: Employment-based opiate abstinence reinforcement
- Opiate Abstinence Reinforcement Only (Experimental): This group would receive employment-based opiate abstinence reinforcement, but this group will not receive VIVITROL.
  Interventions: Behavioral: Employment-based opiate abstinence reinforcement
- Usual Care Control (Other): This group will receive neither abstinence reinforcement nor VIVITROL injections, but they will be invited to attend the workplace and outpatient drug abuse counseling.
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Drug: Vivitrol — Participants receiving this intervention will receive the FDA-approved dose, route, and schedule of administration of VIVITROL. The dose of VIVITROL of 380 mg will be delivered intramuscularly every 4 weeks.
  Arms: VIVITROL&Opiate Abstinence Reinforcement; Vivitrol Only
Behavioral: Employment-based opiate abstinence reinforcement — This intervention will require participants to provide opiate-negative urine samples on Monday, Wednesday and Friday to maintain their maximum pay. If a participant provides an opiate-positive urine sample, or fails to provide a scheduled sample, their base pay will be reset from $8 per hour to $1 per hour. On each day after the reset that the participant provides a urine sample that meets the opiate abstinence criteria and attends the workplace for at least 5 minutes, their base pay will increase by $1 per hour until it reaches the maximum of $8 per hour.
  Arms: Opiate Abstinence Reinforcement Only; VIVITROL&Opiate Abstinence Reinforcement
Other: Usual Care Control — Participants receiving this intervention will be invited to attend the workplace and outpatient drug abuse counseling.
  Arms: Usual Care Control

SUMMARY:
In this 5-year study, the investigators propose to evaluate the separate and combined effects of the FDA-approved formulation of extended release naltrexone (Vivitrol®) and employment-based reinforcement of opiate abstinence in promoting opiate abstinence and reducing risky injection behavior in recently detoxified, opioid-dependent, injection drug users.

DETAILED DESCRIPTION:
Injection heroin use is a chronic problem that fuels the transmission of HIV/AIDS through risky injection behaviors. Methadone and buprenorphine can reduce heroin use and risky injection behavior; however, they have abuse potential, produce physical dependence, can produce lethal overdose, are highly regulated, and some patients simply do not want agonist treatment. Opiate detoxifications can serve as an alternative to agonist treatment, but many injection drug users relapse to heroin use and resume risky injection behaviors after detoxification. Vivitrol®, an extended release formulation of naltrexone, was recently approved by the FDA for the treatment of opioid dependence, but its clinical utility is uncertain given the reluctance of many opioid-dependent adults to maintain its long-term use, and the fact that some patients continue to use opiates while under naltrexone blockade. The investigators research in the first period of this grant showed that employment-based reinforcement can be highly effective in promoting long-term adherence to Vivitrol®. Employment-based reinforcement may be ideally suited to address the limitations of extended release naltrexone by capitalizing on its potential to simultaneously reinforce naltrexone adherence and opiate abstinence. This grant will evaluate the effectiveness of employment-based reinforcement to simultaneously promote high rates of Vivitrol® adherence and increase opiate abstinence. After an opioid detoxification and induction onto oral naltrexone, participants will be invited to attend the Therapeutic Workplace for 24 weeks (where they can work and earn wages) and will be randomly assigned to one of four groups that will differ in whether they receive Vivitrol®, employment-based opiate abstinence reinforcement, both or neither. Participants in Vivitrol® conditions will be required to take scheduled injections to work and earn wages. Participants exposed to opiate abstinence reinforcement will receive a temporary decrease in their workplace pay if they fail to provide an opiate-free urine sample. The study will assess the effects of the interventions on weekly opiate urinalysis results, and on measures of injection drug use and cocaine use. If this study shows that the combined use of Vivitrol® and employment-based reinforcement of adherence and opiate abstinence is effective in maintaining long-term opiate abstinence, this model of employment-based addiction pharmacotherapy could be integrated into community workplaces to disseminate the effective use of Vivitrol®; it could be used to enhance the utility of other new antagonist-like addiction medications; and it could provide an effective means of reducing injection drug use in individuals who persist in injecting heroin and exposing themselves and others to the risk of acquiring or transmitting HIV infection due to their continued injection drug use and risky injection behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. meet the DSM-IV criteria for opioid dependence,
2. report using heroin at least 21 of the last 30 days while living in the community,
3. are unemployed,
4. are 18-65 years old,
5. are medically approved for naltrexone,
6. live in or near Baltimore, MD.

Exclusion Criteria:

1. have current DSM-IV major Axis I disorders
2. have current suicidal or homicidal ideation
3. express interest in methadone treatment
4. are required to use opioids for medical purposes
5. earned over $200 in taxable income over the previous 30 days while living in the community
6. have physical limitations that prevent them from using a keyboard
7. are pregnant or breastfeeding
8. have serum aminotransferase levels over three times normal
9. have known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or poly (lactide-co-glycolide) (PLG) or any other components of the diluents;
10. are participating in any other clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will publish the results in a peer-reviewed journal.

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vivitrol Only | VIVITROL&Opiate Abstinence Reinforcement | Opiate Abstinence Reinforcement Only | Usual Care Control
Started | 25 | 23 | 18 | 18
Completed | 25 | 23 | 18 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vivitrol Only | VIVITROL&Opiate Abstinence Reinforcement | Opiate Abstinence Reinforcement Only | Usual Care Control | Total
Number analyzed (Participants) | 25 | 23 | 18 | 18 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.3) | 43.1 (10.0) | 41.1 (11.1) | 42.2 (11.4) | 42.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 4 | 3 | 24
  Male | 15 | 16 | 14 | 15 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 21 | 13 | 15 | 68
  White | 5 | 2 | 4 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 23 | 18 | 18 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percent of Weekly Urine Samples Negative for Opiates
Description: Was the participant's urine sample negative for opiates at each of the 24 weekly assessments scheduled after random assignment (Y/N)? The outcome measure was the percentage of weekly urine samples that was negative for opiates.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: percentage of negative urine samples
Arm/Group | Vivitrol Only | VIVITROL&Opiate Abstinence Reinforcement | Opiate Abstinence Reinforcement Only | Usual Care Control
Number analyzed (Participants) | 25 | 23 | 18 | 18
percentage of negative urine samples | 64.5 [0 to 100] | 81.3 [0 to 100] | 71.1 [0 to 100] | 66.7 [0 to 100]
Statistical Analysis 1: Comparison: Opiate Abstinence Reinforcement Only vs Usual Care Control; Test type: Superiority; p = 0.48, General Estimating Equation (GEE); Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.2 to 21.6]
Statistical Analysis 2: Comparison: Vivitrol Only vs Usual Care Control; Test type: Superiority; p = 0.61, General Estimating Equation (GEE); Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.1 to 4.6]
Statistical Analysis 3: Comparison: VIVITROL&Opiate Abstinence Reinforcement vs Usual Care Control; Test type: Superiority; p = 0.11, General Estimating Equation (GEE); Odds Ratio (OR) = 6.00, 95% CI 2-sided [0.7 to 54.9]
Statistical Analysis 4: Comparison: VIVITROL&Opiate Abstinence Reinforcement vs Opiate Abstinence Reinforcement Only; Test type: Superiority; p = 0.39, General Estimating Equation (GEE); Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.3 to 24.9]
Statistical Analysis 5: Comparison: Vivitrol Only vs VIVITROL&Opiate Abstinence Reinforcement; Test type: Superiority; p = 0.03, General Estimating Equation (GEE); Odds Ratio (OR) = 10.4, 95% CI 2-sided [1.3 to 85.5]

2. Secondary Outcome: Percent of Weekly Urine Samples Negative for Cocaine
Description: Was the participant's urine sample negative for cocaine at each of the 24 weekly assessments scheduled after random assignment (Y/N)? The outcome measure was the percentage of weekly urine samples that was negative for cocaine.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: percentage of cocaine negative samples
Arm/Group | Vivitrol Only | VIVITROL&Opiate Abstinence Reinforcement | Opiate Abstinence Reinforcement Only | Usual Care Control
Number analyzed (Participants) | 25 | 23 | 18 | 18
percentage of cocaine negative samples | 60.8 [0 to 100] | 68.1 [0 to 100] | 56.3 [0 to 100] | 68.3 [0 to 100]
Statistical Analysis 1: Comparison: Opiate Abstinence Reinforcement Only vs Usual Care Control; Test type: Superiority; p = 0.30, General Estimating Equation (GEE); Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.1 to 2.4]
Statistical Analysis 2: Comparison: Vivitrol Only vs Usual Care Control; Test type: Superiority; p = 0.08, General Estimating Equation (GEE); Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.03 to 1.2]
Statistical Analysis 3: Comparison: VIVITROL&Opiate Abstinence Reinforcement vs Usual Care Control; Test type: Superiority; p = 0.91, General Estimating Equation (GEE); Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.1 to 5.8]
Statistical Analysis 4: Comparison: VIVITROL&Opiate Abstinence Reinforcement vs Opiate Abstinence Reinforcement Only; Test type: Superiority; p = 0.34, General Estimating Equation (GEE); Odds Ratio (OR) = 2.47, 95% CI 2-sided [0.4 to 15.8]
Statistical Analysis 5: Comparison: Vivitrol Only vs VIVITROL&Opiate Abstinence Reinforcement; Test type: Superiority; p = 0.09, General Estimating Equation (GEE); Odds Ratio (OR) = 4.46, 95% CI 2-sided [0.8 to 26.1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vivitrol Only | VIVITROL&Opiate Abstinence Reinforcement | Opiate Abstinence Reinforcement Only | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 1/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/23 | 2/18 | 4/18
Other Adverse Events (participants affected / at risk) | 6/25 | 3/23 | 3/18 | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivitrol Only (N=25) | VIVITROL&Opiate Abstinence Reinforcement (N=23) | Opiate Abstinence Reinforcement Only (N=18) | Usual Care Control (N=18)
death (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The participant never received extended-release naltrexone and all of her urine samples were negative for opiates. At her 6-month follow-up assessment, we were and was told that she had died. The medical examiner believes she had a seizure.
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral menningitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
alcohol detoxification (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychiatric treatment (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weakness on right side of body (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivitrol Only (N=25) | VIVITROL&Opiate Abstinence Reinforcement (N=23) | Opiate Abstinence Reinforcement Only (N=18) | Usual Care Control (N=18)
Abnormal liver function test (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
elbow injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Assault (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Broken ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
leg injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
arm injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychiatric treatment (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver discomfort (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No